CLINICAL TRIAL: NCT03496779
Title: A Phase II Study of Brentuximab Vedotin in Patients With Relapsed or Refractory Peripheral T-cell Lymphoma Treated With Gemcitabine Followed by Brentuximab Vedotin Maintenance
Brief Title: Study of Brentuximab Vedotin in Patients With R/R PTCL Treated With Gemcitabine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TOTAL
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Refractory Peripheral T-Cell Lymphoma; Relapsed Peripheral T-Cell Lymphoma
Keywords: Brentuximab Vedotin; T-cell lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell | interventions — Brentuximab Vedotin; Gemcitabine

STUDY DESIGN:
Intervention Model Description: This study is an open label, multicenter phase 2 study. Patients treated with gemcitabine will receive brentuximab vedotin (GBv) for 4 cycles of induction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Patients treated with gemcitabine will receive Brentuximab Vedotin-induction for 4 cycles of induction.
  Patients who will obtain partial or complete response and who will be eligible for transplant will receive autologous or allogeneic stem cell transplantation.
  Patients who will obtain partial or complete response and who will not be eligible for transplant will receive maintenance therapy with Brentuximab Vedotin-maintenance every 3 weeks for 12 infusions.
  Interventions: Drug: Brentuximab Vedotin - induction; Drug: Gemcitabine; Drug: Brentuximab Vedotin - maintenance; Procedure: autologous or allogeneic stem cell transplantation

INTERVENTIONS:
Drug: Brentuximab Vedotin - induction — Brentuximab vedotin 1.8 mg/kg at D8 of a 28-day cycle - 4 cycles = 16 weeks for combined chemotherapy
  Other Names: Adcetris
Drug: Gemcitabine — Gemcitabine 1000 mg/m² at D1 and D15 of a 28-day cycle - 4 cycles = 16 weeks for combined chemotherapy
  Other Names: Gemzar
Drug: Brentuximab Vedotin - maintenance — Patients who will obtain partial or complete response and who will not be eligible for transplant will receive maintenance therapy with brentuximab vedotin every 3 weeks for 12 infusions.
  Brentuximab vedotin 1.8 mg/kg at D1 of a 21-day cycle - 12 cycles = 36 weeks for maintenance therapy
  Other Names: Adcetris
Procedure: autologous or allogeneic stem cell transplantation — Patients who will obtain partial or complete response and who will be eligible for transplant will receive autologous or allogeneic stem cell transplantation

SUMMARY:
This study is an open label, multicenter phase 2 study. The primary objective of the study is to determine the efficacy of brentuximab vedotin in patients treated by gemcitabine for relapsed or refractory peripheral T-cell lymphoma in term of overall response rate assessed after 4 cycles of treatment according to the international response criteria for malignant lymphoma (Lugano Classification 2014 - CT-Based Response).

DETAILED DESCRIPTION:
Currently, there is no standard treatment for patients with recurrent or refractory peripheral T-cell lymphoma who relapse after a first line of cyclophosphamide, hydroxydaunomycin, oncovin, and prednisone (CHOP) treatment.

Chemotherapies such as gemcitabine are used as monotherapy but the results alone are insufficient. In addition, there is no approved monotherapy in the European Union, with the exception of brentuximab vedotin in refractory or recurrent large systemic anaplastic lymphomas.

Stem cell transplantation may be an option for patients who respond to a second line of treatment or a subsequent line of treatment, but conditions for being eligible for transplantation, including long-term remission, are infrequent.

Brentuximab vedotin (BV) is a targeted treatment directed against a protein, cluster of differentiation antigen 30 (CD30), present on the surface of lymphoma cells. It allows chemotherapy to enter directly into the lymphoma cell. The CD30 protein is variably expressed in patients with relapsed or refractory T-cell lymphoma; about 50% of patients have significant expression.

Data from clinical studies with brentuximab vedotin suggest that the addition of this treatment to gemcitabine may be more successful than gemcitabine alone.

The main hypothesis is a 15% increase in responder patients after 4 cycles of treatment with brentuximab vedotin and gemcitabine. The main objective of the study is therefore to determine the overall response rate after 4 cycles of treatment according to the criteria of Lugano 2014 (response based on CT-scan).

The secondary objectives will focus on the efficacy of brentuximab vedotin: complete response rate, response time for responder patients, time to failure of treatment, time to next treatment and overall survival, efficacy of brentuximab vedotin maintenance: survival progression-free, response time, overall survival, overall response rate based on positron emission tomography (PET)-scan and brentuximab vedotin toxicity in patients treated with gemcitabine and in maintenance therapy.

The duration of the study is estimated to be 4.5 years including follow-up with an estimated recruitment period of 1.5 years. 70 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of 18 years to 80 years of age;
* Understand and voluntarily sign an informed consent document prior to any study related assessment or procedure;
* Patients able to adhere to the study visit schedule and protocol requirements;
* Patients with histologically proven, CD30 positive (at least 5% of cells according to local examination) peripheral T-cell lymphoma (PTCL) according to the 2016 World Health Organization (WHO) classification for whom gemcitabine treatment is expected. A biopsy at relapse is highly recommended;
* Patients who have evidence of relapsed disease after at least one line (and no more than three lines) of treatment or who were refractory to a first or subsequent line of treatment;
* Patients with Ann Arbor stage I - IV;
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2;
* Patients with at least one measurable disease, i.e. one nodal or extra-nodal lesion of 1.5 cm or more;
* Negative pregnancy test for females of childbearing potential (FCBP);
* Female patients of child bearing potential must use an effective method of birth control (i.e. hormonal contraceptive, intrauterine device, diaphragm with spermicide, condom with spermicide or abstinence) during treatment period and 6 months thereafter.
* Males must use an effective method of birth control during treatment period and 6 months thereafter.

Exclusion Criteria:

* Any significant medical condition or laboratory abnormality unrelated to PTCL, or psychiatric illness that would prevent the patient from participating in the study and from signing the informed consent form;
* Any condition that confounds the ability to interpret data from the study;
* Other types of lymphomas, e.g. B-cell lymphoma;
* Central nervous system and/or meningeal involvement by PTCL;
* Signs or symptoms of Progressive Multifocal Leukoencephalopathy;
* Preexistent peripheral neuropathy ≥ grade 2, whatever the cause;
* Contraindication to any drug contained in the chemotherapy regimen;
* Known hypersensitivity to recombinant proteins, murine proteins, or to any excipient contained in the drug formulation of brentuximab vedotin;
* Subjects with HIV or HTLV1 positivity;
* Subjects with active hepatitis B or C. Chronic carriers of hepatitis B without hepatitis B virus (HBV) DNA positive blood are eligible. Subjects with non-active hepatitis C (with normal transaminases) are eligible;
* Chronic or acute, clinically significant, untreated bacterial, viral or fungal infection;
* Any of the following laboratory abnormalities:

  1. Absolute neutrophil count (ANC) < 1500 cells/mm3 (1.5 x 109/L);
  2. Platelet count <75,000/mm3 (75 x 109/L);
  3. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≥ 3.0 x upper limit of normal (ULN). AST or ALT may be elevated up to 5 x ULN if their elevation can be ascribed to the presence of hematologic/solid tumor in the liver;
  4. Serum total bilirubin > 1.5 x ULN;
  5. Serum lipase level > 2 x ULN;
  6. Serum creatinine > 2.0 mg/dL and/or creatinine clearance or calculated creatinine clearance < 40 mL/minute;
  7. Hemoglobin < 8g/dL;
* Active malignancies other than PTCL requiring systemic treatment;
* Previous treatment with brentuximab vedotin;
* Previous treatment with gemcitabine;
* Pregnant or lactating females or women of childbearing potential not willing to use an adequate method of birth control for the duration of the study;
* Known history of any of the following cardiovascular conditions:

  1. Myocardial infarction within 2 years of enrollment
  2. New York Heart Association (NYHA) Class III or IV heart failure
  3. Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
  4. Recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction <50%
* Patients that have not completed any prior treatment chemotherapy and/or other investigational agents within at least 5 half-lives of last dose of that prior treatment;
* Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2018-04-10 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2022-10-08 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | 16 weeks = 4 cycles or permanent treatment discontinuation
  rate of patient in Complete/Partial response according to the international response criteria for malignant lymphoma (Lugano Classification 2014 - CT-Based Response).

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | 16 weeks = 4 cycles or permanent treatment discontinuation
  % of patient who did not progressed according to the international response criteria for malignant lymphoma (Lugano Classification 2014 - CT-Based Response).
Progression-Free Survival (PFS) | 4.5 years
  % of patient who did not progressed according to the international response criteria for malignant lymphoma (Lugano Classification 2014 - CT-Based Response).
Complete Response Rate (CRR) | 16 weeks = 4 cycles or permanent treatment discontinuation
  rate of patient in Complete Response (CR)according to the international response criteria for malignant lymphoma (Lugano Classification 2014 - CT-Based Response).
Duration of Response (DoR) | 16 weeks = 4 cycles or permanent treatment discontinuation
  duration between the Complete/Partial Response and the Progression according to the international response criteria for malignant lymphoma (Lugano Classification 2014 - CT-Based Response) = duration between the Complete/Partial Response and the Progression
Duration of Response (DoR) | 4.5 years
  duration between the Complete/Partial Response and the Progression according to the international response criteria for malignant lymphoma (Lugano Classification 2014 - CT-Based Response) = duration between the Complete/Partial Response and the Progression
Time to Treatment Failure (TTF) | 16 weeks = 4 cycles or permanent treatment discontinuation
  duration between the inclusion and the premature end of treatment
Time to next treatment | 16 weeks = 4 cycles or permanent treatment discontinuation
  Duration between the end of the studied treatment and the beginning of a new one after progression
Overall Survival (OS) | 16 weeks = 4 cycles or permanent treatment discontinuation
  % of patient still alive
Overall Survival (OS) | 4.5 years
  % of patient still alive
Overall response rate | 4.5 years
  rate of patient in Complete/Partial response according to the international response criteria for malignant lymphoma (Lugano Classification 2014 - CT-Based Response).
Number of Serious Adverse Events (SAE) during the induction period | 16 weeks = 4 cycles or permanent treatment discontinuation
Number of Serious Adverse Events (SAE) during the maintenance period | 36 weeks = 12 cycles or permanent treatment discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Richard DELARUE, MD, Study Chair — APHP - Hôpital Necker; Olivier TOURNILHAC, MD, Study Chair — CHU Estaing - Clermont Ferrant
Locations (39):
- Belgium (8):
  - ZNA Stuivenberg, Antwerp
  - A. Z. Sint-Jan, Bruges
  - Clinique Universitaire Saint LUC, Brussels
  - Institut Jules Bordet, Brussels
  - ULB Hôpital Erasme, Brussels
  - UZ Gent, Ghent
  - CHU de Liege, Liège
  - CHU UCL Namur, Yvoir
- France (31):
  - IHBN - CHU Cote de Nacre, Amiens
  - CHU d'Amiens, Amiens
  - CHU Angers, Angers
  - CH d'Avignon - Hôpital Henri Dufaut, Avignon
  - CH Côte Basque, Bayonne
  - CHU de Besançon - Hôpital Jean Minjoz, Besançon
  - CH Chambéry, Chambéry
  - CHU d'Estaing, Clermont-Ferrand
  - APHP - Hopital Henri Mondor, Créteil
  - CHU de Dijon - Hôpital le Bocage, Dijon
  - CHU Grenoble, Grenoble
  - CH de Versailles - Hopital André Mignot, Le Chesnay
  - CH du Mans, Le Mans
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - CHU de Limoges, Limoges
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Annecy Genevois, Metz-Tessy
  - CH Saint-Eloi, Montpellier
  - CH de Mulhouse Sud Alsace, Mulhouse
  - CHU Nancy - Brabois, Nancy
  - CHU de Nantes - Hôtel Dieu, Nantes
  - APHP - Hôpital Necker, Paris
  - APHP - Hôpital Saint Louis, Paris
  - Centre François Magendie - Hôpital du Haut Lévêque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - CHU De Rennes, Rennes
  - Centre Henri BECQUEREL, Rouen
  - CHU de Toulouse, Toulouse
  - CHRU de Tours, Tours
  - CH de Valenciennes, Valenciennes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tournilhac O, Bouabdallah K, Lecolant S, Hacini M, Laribi K, Bailly S, Belmondo T, Maerevoet M, Ysebaert L, Guidez S, Le Gouill S, Bonnet C, Andre M, Dupuis J, Thieblemont C, Bachy E, Daguindau N, Morschhauser F, Tricot S, Moulin C, Banos A, Houot R, Chauchet A, Gyan E, Cartron G, Farhat H, Camus V, Drenou B, Zerazhi H, Sibon D, Nicolas-Virelizier E, Delette C, Snauwaert S, Bailly S, Delarue R, Carras S, Ledoux-Pilon A, Parrens MC, Griolet S, Gaulard P, Delfau-Larue MH, de Leval L, Damaj GL. Brentuximab vedotin addition to gemcitabine in relapsed or refractory peripheral T-cell lymphoma: a LYSA phase 2 study. Blood Adv. 2025 Dec 23;9(24):6292-6304. doi: 10.1182/bloodadvances.2024015787. PMID 40758949
- See also: Website of LYSARC — https://www.lysarc.org/